CLINICAL TRIAL: NCT03586102
Title: Effect of Increased Enteral Protein on Body Composition of Preterm Infants: A Randomized Trial
Brief Title: Effect of Increased Enteral Protein on Body Composition of Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Children's Health System, Alabama (Other)
Responsible Party: Principal Investigator, Ariel A. Salas, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 300000681
Record Dates: First submitted 2018-06-01; First posted 2018-07-13 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Premature Infant
Keywords: Protein supplementation; Human milk fortification
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Clinicians and technicians responsible for the assessment of infant body composition will be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High protein supplementation (Experimental): Infants will receive a diet that consists of mother's own milk or donor human milk and bovine-based human milk fortifier plus a fixed amount of commercially available hydrolyzed bovine protein. The study intervention will begin the day after fortification is ordered and will be continued until postnatal day 50 or 32 weeks postmenstrual age, whichever occurs first.
  Interventions: Dietary Supplement: High protein supplementation
- Standard protein supplementation (Active Comparator): Infants will receive a standard diet that consists of mother's own milk or donor human milk (DHM) and bovine-based human milk fortifier. The study intervention will be continued until postnatal day 50 or 32 weeks postmenstrual age, whichever occurs first.
  Interventions: Dietary Supplement: Standard protein supplementation

INTERVENTIONS:
Dietary Supplement: High protein supplementation — To increase protein content of human milk, a fixed amount of commercially available hydrolyzed bovine protein will be added to fortified human milk. With this pragmatic approach, preterm infants assigned to the high protein supplementation group will receive > 4.5 g/kg/day of enteral protein after establishment of full enteral feeding.
  Arms: High protein supplementation
Dietary Supplement: Standard protein supplementation — Infants assigned to the standard protein supplementation group will receive fortified human milk (< 4.5 g/kg/day of enteral protein)
  Arms: Standard protein supplementation

SUMMARY:
The study hypothesis is that, in human milk-fed extremely preterm infants, higher protein intake compared to usual protein intake reduces percent body fat (%BF) at 3 months of age.

DETAILED DESCRIPTION:
Qualifying participants will be randomly assigned to receive either standard protein supplementation (control group) or high protein supplementation (intervention group).

Intervention group: A fixed amount of commercially available hydrolyzed bovine protein will be added to fortified human milk after establishment of full enteral feeding.

Control group: Hydrolyzed bovine protein will not be added to fortified human milk after establishment of full enteral feeding.

If parent agrees, stool "dirty" diapers will be collected 2 times (at the time of hospital discharge and at 3 months of corrected age).

ELIGIBILITY:
Inclusion Criteria:

* Gestational age between 25 and 28 weeks of gestation
* Feeding volumes of ≥120 ml/kg/day before or on postnatal day 14.

Exclusion Criteria:

* Necrotizing enterocolitis (NEC) stage 2 or greater.
* Gastrointestinal or neurologic malformations.
* Terminal illness needing to limit or withhold support will be exclusion criteria.

Ages: 1 Day to 21 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2018-08-23 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2025-04-24 (Actual)

PRIMARY OUTCOMES:
Infant body composition | Assessed at 36 weeks of postmenstrual age or at 3 months of corrected age
  Percent body fat estimated by air displacement plethysmography

SECONDARY OUTCOMES:
Infant body composition | Assessed at 36 weeks of postmenstrual age or hospital discharge (whichever occurs first)
  Percent body fat estimated by air displacement plethysmography
Growth | Birth to 3 months of corrected age
  Weekly weight gain in grams
Length | Birth to 3 months of corrected age
  Weekly length in cm
Head circumference | Birth to 3 months of corrected age
  Weekly head circumference in cm
Body mass index | Birth to 3 months of corrected age
  Weight and height will be combined to report BMI in kg/m^2
Necrotizing enterocolitis | Postnatal day 14 to postnatal day 120 or discharge, whichever occurs first
  Number of participants with diagnosis of necrotizing enterocolitis stage 2 or 3
Death | Postnatal day 14 to postnatal day 120 or discharge, whichever occurs first

OTHER OUTCOMES:
Changes in intestinal microbiome | Birth to 3 months of corrected age
  Determined by molecular analyses of bacteria in fecal samples
Changes in metabolic pathways | Birth to 3 months of corrected age
  Determined by molecular analyses of serum samples

CONTACTS AND LOCATIONS:
Overall Officials: Ariel A. Salas, MD, MSPH, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Salas AA, Jerome M, Finck A, Razzaghy J, Chandler-Laney P, Carlo WA. Body composition of extremely preterm infants fed protein-enriched, fortified milk: a randomized trial. Pediatr Res. 2022 Apr;91(5):1231-1237. doi: 10.1038/s41390-021-01628-x. Epub 2021 Jun 28. PMID 34183770